CLINICAL TRIAL: NCT04690439
Title: Evaluating the Effectiveness of Photobiomodulation Therapy in the Management of Breast Cancer-Related Lymphedema: a Randomized Controlled Trial
Brief Title: Photobiomodulation Therapy for the Management of Breast Cancer-related Lymphedema
Acronym: LymphLight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-154; B2342020000029 (Registry Identifier: Belgian Registry)
Record Dates: First submitted 2020-12-03; First posted 2020-12-30 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Breast Cancer Related Lymphedema; Lymphedema of Upper Arm
Keywords: Lymphedema; Breast cancer; Photobiomodulation
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema; Lymphedema | interventions — Low-Level Light Therapy; Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: prospective randomized, controlled cross-over trial
Who Masked: Outcomes Assessor
Masking Description: Single : outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will receive first PBM + manual lymphatic drainage for 9 weeks (2 sessions/week), followed by 9 weeks only manual lymphatic drainage.
  Interventions: Device: Photobiomodulation therapy (PBMT); Procedure: Manual Lymphatic drainage
- Group B (Active Comparator): Group B will first receive only manual lymphatic drainage for 9 weeks, followed by the combination of PBM and manual lymphatic drainage for 9 weeks (2x/week).
  Interventions: Device: Photobiomodulation therapy (PBMT); Procedure: Manual Lymphatic drainage

INTERVENTIONS:
Device: Photobiomodulation therapy (PBMT) — The MLS M6 laser from ASA will be used to apply the laser therapy.
  Other Names: LLLT
Procedure: Manual Lymphatic drainage — Patients will receive twice weekly MLT executed by trained physiotherapist
  Other Names: MLT

SUMMARY:
Up to one out of five patients with breast cancer will develop lymphedema in the upper extremity after cancer treatment. Patients with breast cancer-related lymphedema (BCRL) suffer from pain, heaviness, tightness, and a decreased range of motion. Photobiomodulation therapy (PBMT) is a non-invasive therapy based on the application of visible and/or near-infrared light produced by a laser diode or a light-emitting diode. The scientifically proven biologic effects of PBM are improved wound healing, and a reduction in pain, inflammation, and oedema. Therefore, the aim of this study is to evaluate the effectiveness of PBMT on the management of BCRL.

DETAILED DESCRIPTION:
This aim of this study is to determine the efficacy of PBMT in combination with the institutional therapy on the management of BCRL. Therefore, we hypothesize that PBMT in combination with manual lymphatic drainage is able to reduce the limb circumference and the associated pain and improve the QoL of patients with BCRL during treatment and up to 12 months post-treatment.

Primary Objective 1: Arm circumference

The study seeks primarily to determine the effectiveness PBMT and manual lymphatic drainage in reducing the arm circumference in patients with established BCRL during PBM treatment and up to 12 months post-PBMT.

Primary Objective 2: Activity and participation

Another primary aim of this study is to evaluate the effectiveness of PBMT and manual lymphatic drainage in the enhancement of the patients' activity and participation status.

Secondary Objective 1: Pain

A secondary aim of this study is to evaluate if PBMT and manual lymphatic drainage can reduce the BCRL-related pain during PBM treatment and up to 12 months post-PBMT.

Secondary Objective 2: Quality of life

A secondary aim of this study is to evaluate if PBMT and manual lymphatic drainage can improve the patients' QoL during PBM treatment and up to 12 months post-PBMT.

Secondary Objective 3: Depression

A secondary aim of this study is to evaluate if PBMT and manual lymphatic drainage can improve the patients' mental status during PBM treatment and up to 12 months post-PBMT.

Secondary Objective 4: Patient satisfaction

A secondary aim of this study is to evaluate if patients are satisfied with PBMT and manual lymphatic drainage as a treatment for BCRL during the treatment sessions and up to 12 months post-therapy.

Secondary Objective 5: PBM safety

A secondary aim of this study is to evaluate the safety of PBM in oncologic patients up to 5 years post-PBMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Underwent ipsilateral lumpectomy or mastectomy + sentinel lymph node biopsy +/- lymph node dissection
* Underwent radiotherapy with or without chemotherapy
* Diagnosed with BCRL (i.e. International Society of Lymphology (ISL) lymphedema stage I or higher)
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent

Exclusion Criteria:

* Metastatic disease
* Pregnancy
* History of surgery or trauma to the arm
* History of arm infection in the past 3 months
* Use of medications that affect body fluid (e.g., diuretics) in the last 3 months
* Severe psychological disorder or dementia
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Arm circumference and volume | Baseline
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | week 5
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | week 9
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | Week 14
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | Week 18
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | 3 month follow-up
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | 6 month follow-up
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | 9 month follow-up
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm circumference and volume | 12 month follow-up
  The arm circumferences will be measured at olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal of olecranon. The circumference at each point will be recorded in cm.
  The calculated arm volume will be estimated by the formula of the truncated cone of each 4 cm segment proximal (towards the wrist) and distal (towards the acromion) from the olecranon. The following truncated cone formula was used: 4 * (C1* C1 +C1*C2+C2*C2)/12π C1 is the upper circumference and C2 is the lower circumference of each segment. The calculated volume of whole arm is the sum of the volume of all segments of the arm expressed in kubic centimeter
Arm mobility measurement | Baseline
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | week 5
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | week 9
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | week 14
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | week 18
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | 3 month follow-up
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | 6 month follow-up
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | 9 month follow-up
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Arm mobility measurement | 12 month follow-up
  A standard plastic goniometer will be used to measure active range of mobility (ROM) for shoulder flexion, abduction, and external rotation.
Activity and participation | Baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities.
Activity and participation | week 5
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | week 9
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | week 14
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | week 18
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | 3 month follow-up
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | 6 month follow-up
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | 9 month follow-up
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
Activity and participation | 12 month follow-up
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. The score can range from 0 (no disability) to 100 (most severe disability).
ISL classification | Baseline
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | Week 9
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | Week 18
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | 3 month follow-up
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | 6 month follow-up
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | 9 month follow-up
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.
ISL classification | 12 month follow-up
  The severity of BCRL will be evaluated using the ISL criteria. This will be performed by the treating physician.

SECONDARY OUTCOMES:
Pain assessment | Baseline
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | week 5
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | week 9
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | week 14
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | week 18
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | 3 month follow-up
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | 6 month follow-up
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | 9 month follow-up
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Pain assessment | 12 month follow-up
  The patients will be asked to evaluate their pain related to BCRL by using the Visual Analogue Scale (VAS). This scale ranges from 0 (no pain at all) to 10 (extreme agony).
Quality of life assessment | Baseline
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | week 5
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | week 9
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | week 14
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | week 18
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | 3 month follow-up
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | 6 month follow-up
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | 9 month follow-up
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Quality of life assessment | 12 month follow-up
  The validated Lymphedema Functioning, Disability, and Health questionnaire for the upper limb (Lymph-ICF-UL) will be used to evaluate the patients' QoL. This scale ranges from 0 (no problem at all) to 100 (very severe problem).
Depression, anxiety and stress | Baseline
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | week 5
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | week 9
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | week 14
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | week 18
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | 3 month follow-up
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21).
Depression, anxiety and stress | 6 month follow-up
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | 9 month follow-up
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Depression, anxiety and stress | 12 month follow-up
  The mental health of the patients will be determined using the Depression Anxiety Stress-Scale (DASS-21). Three different scores will be calculated: depression (0-21), anxiety (0-21) and stress (0-18). A lower score indicates a normal mental health, while a higher score indicates extremely severe depression, anxiety and/or stress.
Patients' satisfaction with the therapeutic intervention | At week 9
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patients' satisfaction with the therapeutic intervention | At week 18
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patients' satisfaction with the therapeutic intervention | 3 month follow-up
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patients' satisfaction with the therapeutic intervention | 6 month follow-up
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patients' satisfaction with the therapeutic intervention | 9 month follow-up
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patients' satisfaction with the therapeutic intervention | 12 month follow-up
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention and their global satisfaction with the therapeutic intervention, using the Numerical Rating Scale (NRS). This is scored on a scale from 0 (extremely dissatisfied) to 10 (extremely satisfied).

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | 3 month follow-up
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | 6 month follow-up
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | 9 month follow-up
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | 12 month follow-up
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
Appearance and date of local and regional recurrence | 12 month follow-up
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 2 years follow up
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 3 years follow up
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 4 years follow up
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 5 years follow up
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of secondary tumors | 1 year follow up
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 2 years follow up
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 3 years follow up
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 4 years follow up
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 5 years follow up
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of distant metastasis | 1 year follow up
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 2 years follow up
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 3 years follow up
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 4 years follow up
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 5 years follow up
  The possible appearance and date of distant metastasis will be collected.
Date of death of any cause | 1 year follow up
  If the patient dies within the first year after the treatment, their date of death will be collected.
Date of death of any cause | 2 years follow up
  If the patient dies within 2 years after the treatment, their date of death will be collected.
Date of death of any cause | 3 years post treatment
  If the patient dies within 3 years after the treatment, their date of death will be collected.
Date of death of any cause | 4 years follow up
  If the patient dies within 4 years after the treatment, their date of death will be collected.
Date of death of any cause | 5 years follow up
  If the patient dies within 5 years after the treatment, their date of death will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Jessa Hospital
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No